CLINICAL TRIAL: NCT04774120
Title: Relationship Between Bispectral Index, EEG Features, and Propofol Effect-site Concentration in Young and Elderly Patients.
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 200726002
Record Dates: First submitted 2021-01-19; First posted 2021-03-01 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-02

CONDITIONS: Electroencephalography; Aging; Propofol; Depth of Anesthesia
Keywords: electroencephalography; bispectral index; propofol; alpha band; aging; burst suppression
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Young Patients (Patients aged 18 to 65 years.): Propofol infusion rate will be started at 20-25 mg/kg/hr until SR achieved. Then restarted at half of the initial rate. Maintenance of anesthesia will be guided by Sedline Monitor to maintain an alpha band present in the spectrogram and SEF95 between 8-12 Hz. BIS monitor will be covered. Both EEG signals (Sedline and BIS) will be registered simultaneously until the patient's extubation.
  Interventions: Drug: Propofol
- Elderly patients (Patients aged 65 to 85 years. ): Propofol infusion rate will be started at 15-20 mg/kg/hr until SR achieved. Then restarted at half of the initial rate. Maintenance of anesthesia will be guided by Sedline Monitor to maintain an alpha band present in the spectrogram and SEF95 between 8-12 Hz. BIS monitor will be covered. Both EEG signals (Sedline and BIS) will be registered simultaneously until the patient's extubation.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol will be started at a rate of 15-20 mg/kg/hr in patients >65 years and 20-25 mg/kg/hr in younger patients (<65 years) until a suppression rate (SR) is achieved. If not, can be increased by 5 mg/kg/hr every 5 minutes up to 25 mg/kg/hr in the elderly group and 30 mg/kg/hr in the younger group or after 15 minutes have passed. When the SR appears, propofol infusion will be stopped. Then restarted at half of the initial rate. Maintenance of anesthesia will be guided by Sedline Monitor to maintain an alpha band present in the spectrogram and SEF95 between 8-12 Hz. BIS monitor will be covered. Both EEG signals (Sedline and BIS) will be registered simultaneously until the patient's extubation.
  Other Names: Diprivan; Propoven

SUMMARY:
The aim of this study is to describe the BIS values and electroencephalographic patterns during total intravenous anesthesia with propofol-remifentanyl, in patients from 18 to 85 years.

DETAILED DESCRIPTION:
Propofol is an anesthetic drug regularly used in elderly patients requiring anesthesia. The electroencephalographic pattern recognized when propofol is administered is different from the pattern obtained in younger patients. Both groups present alpha and slow delta bands, but younger patients present more intense electroencephalographic bands than older patients (1). The correlation between BIS values and the power of electroencephalographic frequency bands during propofol-remifentanyl anesthesia has not been determined.

The investigators will describe the changes in BIS values and electroencephalographic patterns in young and elderly patients receiving propofol-remifentanyl anesthesia for elective surgery, at different propofol concentration levels. Formal characterization of the dynamic relationship between propofol concentrations at the effect site (Ce), spectral power, and BIS values may provide clinically relevant information to design propofol dose schemes in elderly patients.

The investigators will carry out a prospective observational clinical study at the Clinical Hospital of the Catholic University of Chile. 30 patients, aged 18-85 years, scheduled to undergo elective surgery will be recruited. Standard monitoring and 2 frontal EEG monitors will be installed: Sedline® and BIS®. The electroencephalographic signal from these monitors will be recorded simultaneously from anesthesia induction until extubation. Propofol will be started at a rate of 15-20 mg/kg/hr in patients >65 years and 20-25 mg/kg/hr in younger patients (<65 years) until a suppression rate (SR) >1% appears in the BIS® EEG monitor. If the SR is not achieved, the infusion rate can be increased by 5 mg/kg/hr every 5 minutes until 25 mg/kg/hr in the elderly group and 30 mg/kg/hr in the younger group. When the SR appears, propofol infusion will be stopped. The induction phase will be considered completed at this point. Loss of response (LOR), defined as the timepoint when patients became unresponsive to verbal commands, soft shaking, and eyelash reflex, will be assessed every 30 seconds. When patients become apneic, positive pressure mask ventilation will be started gently at a rate of 10 breaths per minute. After induction of anesthesia, opioids and neuromuscular blocking drugs will be given to facilitate tracheal intubation. When BIS values increase to recommended hypnotic levels for surgery (40-60), the propofol infusion rate will be started again at half of the induction rate. This rate will be adjusted to maintain the alpha band present in the Sedline spectrogram and SEF95 between 8-12 Hz. BIS monitor will be covered and hidden from the attending anesthesiologist during the maintenance phase. After surgery ends, EEG monitoring will continue until the patient's extubation. One hour after extubation, the Brice questionnaire will be performed to detect intraoperative awakening. Propofol concentration will be estimated using the Schnider model.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective surgery requiring general anesthesia.
* American Society of Anesthesiology (ASA) Score I or II

Exclusion Criteria:

* Patients with neurological diseases or history of cognitive impairment.
* Requiring the use of two or more drugs affecting Central nervous system
* History of drugs or alcohol abuse
* Body mass index over 35 kg/m^2
* Propofol allergy
* Cardiac congestive failure
* History of coronary syndrome

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly patients scheduled for surgery are an understudied population. Incidence of postoperative delirium and other complications can be related to changes in cerebral dynamics under anesthesia, with effects observed even after the use of anesthetics agents.
  Formal characterization of the dynamic relationship between propofol concentrations at the effect site (Ce), spectral power, and BIS values may provide clinically relevant information to design propofol dose schemes in young and elderly patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
BIS values at which EEG patterns appears during induction of anesthesia with propofol. | From induction of anesthesia until suppression rate appears, an average of 15 minutes.
  BIS values correlated to specific EEG patterns (frequency bands, complexity measures and burst suppression)

SECONDARY OUTCOMES:
Propofol effect-site concentration (µg/ml) required to observe specific EEG patterns | From induction of anesthesia until loss of consciousness, an average of 15 minutes.
  Propofol effect-site concentrations achieved at the time that specific EEG patterns appear (frequency bands power, complexity measures and burst suppression).
Propofol effect-site concentration (µg/ml) required to achieve loss of consciousness | From Induction of anesthesia until suppression rate appears, an average of 15 minutes.
  Propofol effect-site concentration (µg/ml) at the moment of loss of consciousness
BIS values at loss of consciousness | From Induction of anesthesia until suppression rate appears, an average of 15 minutes.
  BIS values at the moment of loss of consciousness
Percentage of time with BIS values between 40-60 and out of this range. | From induction of anesthesia until patient's extubation, an average of 90 minutes.
  Percentage of time that BIS values are between 40-60 and out of this range.
Time to achieve loss of consciousness | From Induction of anesthesia until loss of consciousness, an average of 10 minutes.
  Time (minutes) to achieve loss of consciousness.
Time to achieve loss suppression rate >1% in BIS monitor. | From Induction of anesthesia until suppression rate appears, an average of 15 minutes.
  Time (minutes) to achieve loss suppression rate >1% in BIS monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Muñoz, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Division de Anestesia - Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Purdon PL, Pavone KJ, Akeju O, Smith AC, Sampson AL, Lee J, Zhou DW, Solt K, Brown EN. The Ageing Brain: Age-dependent changes in the electroencephalogram during propofol and sevoflurane general anaesthesia. Br J Anaesth. 2015 Jul;115 Suppl 1(Suppl 1):i46-i57. doi: 10.1093/bja/aev213. PMID 26174300